CLINICAL TRIAL: NCT06529354
Title: The Role of Exercise Intensity in Water Aerobics: Improving Health Markers in Adults and Older Adults Over 24 Weeks
Brief Title: 24-Week Water Aerobics Program for Adults and Older Adults at Different Intensity Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beira Interior (Other)
Responsible Party: Principal Investigator, Luís Oliveira Brandão Faíl, Principal Investigator, University of Beira Interior
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CE-UBI-Pj-2019-051
Record Dates: First submitted 2024-07-15; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Aquatic exercise; Intensity; Physical fitness; Health-related; Quality of life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-intensity Group (Experimental): Participants engaged in 45-minute water aerobics sessions twice a week for 24 weeks at moderate intensities.
  Interventions: Behavioral: Moderate-intensity Group
- High-intensity Group (Experimental): Participants engaged in 45-minute water aerobics sessions twice a week for 24 weeks at high intensities.
  Interventions: Behavioral: High-intensity Group

INTERVENTIONS:
Behavioral: Moderate-intensity Group — In water aerobics sessions, the exercises are performed at a moderate intensity, between 60% and 70% of the participant's maximum heart rate predicted by their age.
  Arms: Moderate-intensity Group
Behavioral: High-intensity Group — In water aerobics sessions, the exercises are performed at a high intensity, between 80% and 90% of the participant's maximum heart rate predicted by their age.
  Arms: High-intensity Group

SUMMARY:
This goal of this clinical trial is to verify the best way to do water aerobics with adults and older adults. It wants to answer these questions:

* Is high-intensity water aerobics better than water aerobics performed at moderate intensity?
* Does a 24-week water aerobics program improve muscle strength, body weight, fat mass, triglycerides, cholesterol, blood pressure, and quality of life for adults and older adults?

Participants must:

* Do water aerobics at high or moderate intensity, twice a week for 45 minutes per class, for 24 weeks.
* Be assessed before starting the water aerobics program and after it ends to see if there are gains in muscle strength, body weight, fat mass, triglycerides, cholesterol, blood pressure, and quality of life.

It was believed that all variables would get better after doing water aerobics, no matter the intensity. It was also expected that doing higher-intensity water aerobics would lead to larger gains in all measurements compared to moderate-intensity.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age

Exclusion Criteria:

* taking part in another physical exercise program
* being recently hospitalized
* having severe motor or cognitive problems
* having any medical restrictions on physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in explosive strength of lower limbs at 24 weeks | Baseline and week 25
  The countermovement jump was used to assess the explosive strength of the lower limbs. Participants were instructed to perform three countermovement jumps, aiming to jump as high as possible, with one minute of rest between each jump. A higher jump height indicates a better score in this evaluation. The mean value of the three jumps was considered for the test.
Change from Baseline in explosive strength of upper limbs at 24 weeks | Baseline and week 25
  The explosive strength of the upper limbs was measured by having participants throw a 3-kilogram medicine ball, with the best scores achieved by throwing the ball as far as possible. Three throws were performed, and the mean value was used in this test.
Change from Baseline in endurance strength of lower limbs at 24 weeks | Baseline and week 25
  The chair stand test was used to evaluate the endurance strength of the lower limbs. Participants sat in the center of a chair with a straight back and feet shoulder-width apart and in full contact with the floor. They then rose to maximum extension and returned to the initial sitting position, aiming to complete as many repetitions as possible within a 30-second.
Change from Baseline in endurance strength of upper limbs at 24 weeks | Baseline and week 25
  The arm curl test assessed the upper limbs' endurance strength. Participants were seated in a chair with a straight back and their feet flat on the floor, holding a 2 kg dumbbell in their dominant hand. They were instructed to perform as many correct flexions as possible within a 30-second time limit.
Change from Baseline in body mass at 24 weeks | Baseline and week 25
  A bioimpedance balance was used for this test, with participants being barefoot and dressed in minimal clothing.
Change from Baseline in fat mass percentage at 24 weeks | Baseline and week 25
Change from Baseline in fat-free mass at 24 weeks | Baseline and week 25
Change from Baseline in body mass index at 24 weeks | Baseline and week 25
  The body mass index (BMI) was calculated by dividing the body mass value by the height squared (kg/m^2). For this, each participant's height was measured using a precision stadiometer with a scale of 0.001 m. For the correct extraction of this test, participants were barefoot.
Change from Baseline in triglycerides at 24 weeks | Baseline and week 25
  Blood samples were collected before exercise (after a 15-minute rest period) and at least 2 hours after the last meal.
Change from Baseline in total cholesterol at 24 weeks | Baseline and week 25
Change from Baseline in diastolic blood pressure at 24 weeks | Baseline and week 25
  The automatic blood pressure monitor was used to measure the participants' blood pressure after seated and rested for 20 minutes.
Change from Baseline in systolic blood pressure at 24 weeks | Baseline and week 25
Change from Baseline in resting heart rate at 24 weeks | Baseline and week 25
  Resting heart rate was assessed using an automatic blood pressure monitor, after the participant was seated and resting for at least 20 minutes.

SECONDARY OUTCOMES:
Change from Baseline in quality of life at 24 weeks | Baseline and week 25
  The WHOQOL-BREF (Portuguese version) questionnaire, consisting of 26 items, was used to evaluate the participants' quality of life. Of the 26 items, 2 pertain to general quality of life and general health, while the remaining 24 items assess the perception of quality of life in 4 domains: physical, psychological, social relationships, and environment. Higher scores indicate a higher quality of life in each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Luís Faíl, Principal Investigator — University of Beira Interior
Locations (1):
- Tramagal Municipal Swimming Pool, Abrantes, Portugal

IPD SHARING:
Plan to Share IPD: No